CLINICAL TRIAL: NCT04023188
Title: CART Phase 2 Study: Diagnostic Performance of a Ring-type Wearable Device Using Deep Learning Analysis of Photoplethysmographic Signals for Detecting Atrial Fibrillation
Brief Title: A Ring-type Wearable Device for Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Sky Labs Inc. (Unknown)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Other Study IDs: CART2
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; deep learning; diagnosis; photoplethysmography; wearable electronic devices
MeSH Terms: conditions — Atrial Fibrillation; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates diagnostic performance of a ring-type wearable device for detecting atrial fibrillation. This is a prospective cohort registry study began after the date of IRB approval and until 31th Dec. 2019. The eligible criteria are (1) those who admitted the institution for elective direct-current cardioversion of persistent atrial fibrillation, and (2) aged 19 years or more. The exclusion criteria are (1) those aged less than 19 years, (2) those who are not eligible to perform cardioversion by any reasons. This study aims to recruit 200 participants in total. The participants are required to record photoplethysmographic signals by the ring device in addition to routine procedures of direct-current cardioversion, hence, the study is at minimal risk.

DETAILED DESCRIPTION:
1. Study title: Diagnostic Performance of a Ring-type Wearable Device Using Deep Learning Analysis of Photoplethysmographic Signals for Detecting Atrial Fibrillation.
2. Study type: Investigator initiated study.
3. Study design: Prospective observational cohort registry design.
4. Sponsor: Sky Labs, Inc., Republic of Korea.
5. The aim of the study: To evaluate diagnostic performance of a ring-type wearable device for detecting atrial fibrillation.
6. Study period: From the date of IRB approval to 31th Dec. 2019.
7. The size of study population: 200 participants
8. The eligibility criteria:

(1) Those with persistent atrial fibrillation (2) Those who admitted the institution for elective direct-current cardioversion (3) Those aged 19 years or more 9. The exclusion criteria:

(1) Those with other forms of cardiac arrhythmias (2) Those aged less than 19 hears (3) Those who are not eligible to perform electrical cardioversion 10. Procedures of the study

1. A participant is under the routine procedures of direct-current cardioversion.
2. On admission, a participant is given with detailed information of the study.
3. After the informed consent, the only additional procedure due to the study is recording photoplethysmographic signal by wearing a ring-type device.
4. Recorded signals are evaluated without encompassing persornal information. 11. Financial benefits to the participants: None.

ELIGIBILITY:
Inclusion Criteria:

* Those with persistent atrial fibrillation
* Those who admitted for elective direct-current cardioversion
* Those who aged 19 years or more

Exclusion Criteria:

* Those who aged less than 19 years
* Those who had other types of cardiac arrhythmias
* Those who are not eligible to perform electrical cardioversion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study consecutively recruits participants who admitted for elective direct-current cardioversion due to persistent atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | Baseline
  Diagnostic performance of a ring-type wearable device for detecting atrial fibrillation (parameters including sensitivity, specificity, positive predictive value, negative predictive value).

CONTACTS AND LOCATIONS:
Overall Officials: Eue-Keun Choi, MD, PhD, Principal Investigator — Devision of Cardiology, Department of Internal Medicine, Seoul National University Hospital
Locations (1):
- Seoul National university Hostpital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Currently, according to the decision with IRB of the institution, the IPD is not planned to be shared with other researchers for the purpose of protecting potential privacy issues of the participants.

REFERENCES:
- [Derived] Kwon S, Hong J, Choi EK, Lee B, Baik C, Lee E, Jeong ER, Koo BK, Oh S, Yi Y. Detection of Atrial Fibrillation Using a Ring-Type Wearable Device (CardioTracker) and Deep Learning Analysis of Photoplethysmography Signals: Prospective Observational Proof-of-Concept Study. J Med Internet Res. 2020 May 21;22(5):e16443. doi: 10.2196/16443. PMID 32348254